CLINICAL TRIAL: NCT04605172
Title: The Impact of the SARS CoV-2 Lockdown Policy on Spontaneous Premature Birth at the Regional University Maternity Hospital of Nancy
Brief Title: Lockdown Impact on Spontaneous Premature Birth in a Level III NICU
Acronym: CONFINéo
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jean-Michel HASCOET, Professor, Central Hospital, Nancy, France
Other Study IDs: 2020PI168
Record Dates: First submitted 2020-10-22; First posted 2020-10-27 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Premature Birth; Preterm Labor
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature | interventions — Hospitalization

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lockdown Group: newborn born prematurely during confinement (1st March - 1st June 2020)
  Interventions: Other: hospitalization for premature birth
- Control group: newborn born prematurely in comparative years over the same period (1st March - 1st June from 2015 to 2019)
  Interventions: Other: hospitalization for premature birth

INTERVENTIONS:
Other: hospitalization for premature birth — Number of inborn and outborn infants prematurely born during a specific period of time

SUMMARY:
Preterm labor (PL) is the leading cause of hospitalization during pregnancy and premature birth the leading cause of fetal morbidity and mortality in France. PL is defined by regular and painful uterine contractions associated with a change in the cervix, between 22 and 36 weeks of gestation.

It has been shown that the risk of spontaneous prematurity increases particularly in case of working over 40 hours per week, hard physically conditions, or prolonged daily transport time. Rest is one of the most efficient measure to prevent PL and should be proposed to all pregnant women, and combined with other therapies such as tocolysis or cerclage when needed.

The very particular period of lockdown during the COVID-19 pandemic had pregnant women to drastically reduce their activity. They suspended their work and stayed home for various reasons such as pregnancy in progress, children at home, and also collective reasons such as teleworking or workplace closure.

During the lockdown period from March 17th to May 11th 2020, fewer preterm labor and less spontaneous prematurity have been suspected by the neonatology and obstetrics teams throughout the Lorraine region.

Our study aims to objectively confirm this observation. In this investigation we aim to find a relationship between lockdown, PL and spontaneous prematurity which would need to re-evaluate public health recommendations for pregnant women outside the lockdown.

ELIGIBILITY:
Inclusion Criteria:

* Any prematurely born infant before 37 SA and care for by the level III NICU, over the predefined periods.

Exclusion Criteria:

* non premature newborn

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All premature newborns born before 37 SA and care for by the level III NICU of the Maternité Régionale Universitaire de Nancy, over time periods from March 1 to June 1 of the years 2015 to 2020.
Sampling Method: Non-Probability Sample
Enrollment: 812 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the impact of confinement on the rate of spontaneous prematurity at the Regional University Maternity Hospital of Nancy (MRUN) | baseline
  Number of prematurely born infants

SECONDARY OUTCOMES:
Evaluate the impact of confinement on the type of prematurity rate: spontaneous or not | baseline
  Number of infants born by vaginal delivery or cesarean section
Evaluate the impact of confinement on the outborn rate managed by the Regional Neonatal transport team for prematurity | baseline
  Number of infants transferred from referring hospitals to the level III NICU for prematurity
Evaluate the type of prematurity over the period of confinement | baseline
  Diagnosis evaluation of prematurely born infants during lockdown period

CONTACTS AND LOCATIONS:
Locations (1):
- Maternite Regionale Universitaire CHRU NANCY, Nancy, Lorraine, France